CLINICAL TRIAL: NCT04498962
Title: The Effect of Danzhu Fuyuan Granule as Adjunctive Therapy for Chronic Stable Angina, Vascular Dementia and Idiopathic Membranous Nephropathy: A Bayesian Basket Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jingqing Hu (Other)
Responsible Party: Sponsor-Investigator, Jingqing Hu, Director of Institute of Basic Theory of Traditional Chinese Medicine, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019YFC1708500
Record Dates: First submitted 2020-07-21; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Chronic Stable Angina; Vascular Dementia; Idiopathic Membranous Nephropathy
Keywords: Danzhu Fuyuan Granule; Basket Trial
MeSH Terms: conditions — Angina, Stable; Dementia, Vascular; Glomerulonephritis, Membranous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- chronic stable angina (Experimental): Experimental: the patient who have the syndrome of intermingled phlegm and blood stasis with chronic stable angina will be treated by Danzhu Fuyuan Granule in addtion to routine care
  Interventions: Drug: Danzhu Fuyuan Granule
- Vascular Dementia (Experimental): Experimental: the patient who have the syndrome of intermingled phlegm and blood stasis with Vascular Dementia will be treated by Danzhu Fuyuan Granule in addtion to routine care
  Interventions: Drug: Danzhu Fuyuan Granule
- Idiopathic Membranous Nephropathy (Experimental): Experimental: the patient who have the syndrome of intermingled phlegm and blood stasis with Idiopathic Membranous Nephropathy will be treated by Danzhu Fuyuan Granule in addtion to routine care
  Interventions: Drug: Danzhu Fuyuan Granule
- Healthy population (No Intervention): Comparator: Healthy population with no treatment

INTERVENTIONS:
Drug: Danzhu Fuyuan Granule — Danzhu Fuyuan Granules，2 times / day, 1 bag / time, one time in the morning and one time in the evening. It is recommended to add the same amount of boiling water as the particles to soak for 30 seconds, and then add 5 times boiling water to dissolve until completely dissolved.The treatment cycle of each arm: 8 weeks for Chronic Stable Angina, 6 months for Vascular Dementia and 6 months for Idiopathic Membranous Nephropathy.
  Arms: Idiopathic Membranous Nephropathy; Vascular Dementia; chronic stable angina

SUMMARY:
This study is designed as a bayesian basket trial , which aims to evaluate the efficacy of Danzhu Fuyuan Granule in patients with Chronic Stable Angina, Vascular Dementia and Idiopathic Membranous Nephropathy

ELIGIBILITY:
Eligibility Criteria for Chronic Stable Angina group

Inclusion criteria for Chronic Stable Angina group

1. Patient must be between the ages of 40 and 70 years
2. Evidence of coronary artery disease that consists of a well-documented medical history (over 3 months prior to the enrollment) of myocardial infarction or significant coronary artery disease with noninvasive or angiographic confirmation.
3. Patient must match the diagnostic criteria for chronic stable angina set by Chinese Medical Association;
4. The number of angina pectoris attacked in the past 3 months was more than 2 times per week
5. Class I or Class II, Grading of Angina Pectoris by the Canadian Cardiovascular Society Classification System
6. Patients who met the clinical diagnostic criteria for Syndrome of intermingled phlegm and blood stasis with chronic stable angina;
7. The results of Treadmill Exercise Test were positive;
8. All other Traditional Chinese Medicine interventions (including decoction, granule, proprietary Chinese medicine, acupuncture, etc.) should be stopped for 2 weeks or more;
9. They signed the consent form voluntarily and agreed to participate in the research.

Exclusion criteria for Chronic Stable Angina group

1. patients who are diagnosed with acute coronary syndrome (including acute myocardial infarction or unstable angina pectoris) occurred within 2 months before enrollment, or had undergone revascularization within 3 months before enrollment, or planned to undergo revascularization during the study period;
2. Patients who are unable to complete Treadmill Exercise Test for various reasons, including absolute and relative contraindications;
3. Severe primary diseases such as respiratory, blood system or malignant tumor, or known renal insufficiency (serum creatinine (CR) > 221 umol /L in male, or 177 umol / L in female);
4. Patients with epilepsy who had bleeding tendency, history of cerebral hemorrhage, or needed anticonvulsant therapy;
5. Patients with active liver disease, or accompanied with unexplained continuous increase of serum transaminase, or the detection value of alanine aminotransferase (ALT) and aspartate aminotransferase (AST) is more than twice the upper limit of normal reference value;
6. Pregnancy or lactation;
7. patients can't stopped taking long-acting nitrates during the clinical trial;
8. undergoing other clinical trials;
9. There was a history of alcoholism or drug dependence in the past two years;
10. Other situations that the research physician thinks are not suitable to participate in this trial include but are not limited to: the subjects cannot follow the research protocol, which will bring potential safety hazards to the subjects, etc.

Eligibility Criteria for Vascular Dementia group

Inclusion criteria for Vascular Dementia group

1. The age of the subjects was 35-85 years old;
2. It was in accordance with the diagnostic standard of Western medicine for vascular dementia;
3. It is in accordance with the diagnostic standard of TCM phlegm and blood stasis syndrome of vascular dementia;
4. They signed informed consent and volunteered to participate in the study;
5. The patients are expected to follow up within half a year.

Exclusion criteria for vascular dementia group

1. Early memory impairment with progressive deterioration, early prominent features of Parkinson's disease, and primary nervous system diseases (such as multiple sclerosis, encephalitis, etc.);
2. There was no vascular lesion in neuroimaging examination;
3. Other diseases that can explain cognitive impairment, such as brain tumor, multiple sclerosis, encephalitis, depression, poisoning, and systemic diseases and metabolic abnormalities that significantly affect cognitive function;
4. Severe heart, brain, liver and hematopoiesis diseases, or other serious diseases affecting their survival;
5. Drug or alcohol abuse / dependence within 3 months before participating in the trial;
6. Pregnant and lactating women;
7. Patients with severe mental disorders (perception disorders, thinking disorders);
8. For known renal insufficiency, serum creatinine (CR) was higher than 221 umol/L in male and 177 umol/L in female;
9. Patients with known liver dysfunction, alanine aminotransferase (ALT) > 3 times of normal value or with cirrhosis;
10. The researchers believe that there are other situations that are not suitable for participating in this study.

Eligibility Criteria for Idiopathic Membranous Nephropathy group

Inclusion criteria for Idiopathic Membranous Nephropathy group

1. The pathological diagnosis of renal biopsy was membranous nephropathy;
2. The syndrome of TCM is phlegm and blood stasis;
3. The urinary protein was more than 1G / D and < 8g / d;
4. Blood pressure can be effectively controlled at ≤ 140 / 90mmHg;
5. eGFR≥45ml/min；
6. The age ranged from 18 to 70 years old;
7. Sign informed consent.

Exclusion criteria for Idiopathic Membranous Nephropathy group

1. All kinds of secondary membranous nephropathy;
2. Those who are taking hormone and / or immunosuppressive therapy;
3. Women with pregnancy planning, pregnancy and lactation;
4. Severe heart, brain, liver and hematopoiesis diseases, or other serious diseases affecting their survival;
5. Participants in other clinical trials in recent 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint 1 for Chronic Stable Angina Group: the time to ST depression at the end of week 8 compared with baseline on submaximal exercise Modified Bruce Protocol | 8 weeks
  It is suitable for Chronic Stable Angina group. The time to ST depression at the end of week 8 compared with baseline on submaximal exercise Modified Bruce Protocol
Primary endpoint 2 for Chronic Stable Angina group: the score on Syndrome Questionnaire of Intermingled Phlegm and Blood Stasis with Chronic Stable Angina at the end of week 8 compared with baseline | 8 weeks
  It is suitable for Chronic Stable Angina group. Syndrome Questionnaire of Intermingled Phlegm and Blood Stasis with Chronic Stable Angina is a questionnarie to evaluate the severity of Syndrome of Intermingled Phlegm and Blood Stasis with Chronic Stable Angina. The minimum score is 0 and the maximum score is 41. The higher the score is, the worse the outcomes is.
Primary endpoint 1 for Vascular Dementia group: the score of Mini-mental State Examination at the end of month 6 compared with baseline | 6 month
  It is suitable for Vascular Dementia group. Mini Mental State Examination gives the 'mini-mental state' examination of cognitive function. This is a 5-minute bedside test that is useful as a screen and in assessing the degree of cognitive dysfunction in patients with diffuse brain disorders. The minimum score is 0 and the maximum score is 30. The higher the score is, the better the outcomes is.
Primary endpoint 2 for Vascular Dementia group: the score on Syndrome Questionnaire of Intermingled Phlegm and Blood Stasis with Vascular Dementia at the end of month 6 compared with baseline | 6 month
  It is suitable for Vascular Dementia group Syndrome Questionnaire of Intermingled Phlegm and Blood Stasis with Vascular Dementia is a questionnarie to evaluate the severity of Syndrome of Intermingled Phlegm and Blood Stasis with Vascular Dementia. The minimum score is 0 and the maximum score is 46. The higher the score is, the worse the outcomes is.
Primary endpoint 1 for Idiopathic Membranous Nephropathy group: level of the 24 hour urine protein quantification at the end of month 6 compared with baseline | 6 months
  It is suitable for Idiopathic Membranous Nephropathy group. level of the 24 hour urine protein quantification at the end of month 6 compared with baseline. To evaluate the drug efficiency by comparing date changes of 24 hour urine protein quantification before and 6 months after treatment by Danzhu Fuyuan Granule . The unit of 24 hour urine protein quantification values is described as g/24h
Primary endpoint 2 for Idiopathic Membranous Nephropathy group: the score on Syndrome Questionnaire of Intermingled Phlegm and Blood Stasis with Idiopathic Membranous Nephropathy at the end of month 6 compared with baseline | 6 months
  It is suitable for Idiopathic Membranous Nephropathy group. Syndrome Questionnaire of Intermingled Phlegm and Blood Stasis withIdiopathic Membranous Nephropathy is a questionnarie to evaluate the severity of Syndrome of Intermingled Phlegm and Blood Stasis with Idiopathic Membranous Nephropathy. The minimum score is 0 and the maximum score is 42. The higher the score is, the worse the outcomes is.

SECONDARY OUTCOMES:
Duke treadmill score (DTS) at the end of week 8 compared with baseline on submaximal exercise Modified Bruce Protocol | 8 weeks
  It is suitable for Chronic Stable Angina group. The Duke Treadmill Score was introduced in 1991 as a set of treadmill exercise findings that predict individual risk for death on the basis of a weighted combination of exercise duration, ST-segment depression, and the presence and nature of angina during testing. The score is calculated by subtracting 5 times the ST depression (in millimeters) and 4 times the angina score (no angina = 0, nonlimiting angina = 1, and test-limiting angina = 2) from minutes of exercise duration on the Modified Bruce protocol
the score on Seattle Angina Questionnaire | 8 weeks
  It is suitable for Chronic Stable Angina group. The Seattle Angina Questionnaire (SAQ) is a self-administered, disease-specific measure for patients with Cornary Artery Disease that is valid, reproducible, and sensitive to clinical change.
  The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Each scale is transformed to a score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life).
Frequency of weekly angina episodes | 8 weeks
  It is suitable for Chronic Stable Angina group
Angina pectoris severity classification according to Canadian Cardiovascular Society (CCS) | 8 weeks
  It is suitable for Chronic Stable Angina group
Stopping or reducing rate of the Nitroglycerin Table | 8 weeks
  It issuitable for Chronic Stable Angina group
Number of subjects with adverse events or severe adverse events | 8 weeks
  It is suitable for Chronic Stable Angina group
Brain pulse index mearsured by Transcranial Doppler | 6 months
  It is suitable for Vascular Dementia group
Arterial systolic blood flow velocity mearsured by Transcranial Doppler | 6 months
  It is suitable for Vascular Dementia group
Mean flow velocity mearsured by Transcranial Doppler | 6 months
  It is suitable for Vascular Dementia group
Level of serum creatinine | 6 months
  It is suitable for Idiopathic Membranous Nephropathy group.
Level of blood urea nitrogen | 6 months
  It is sutitable for Idiopathic Membranous Nephropathy group.
Glomerular filtration rate | 6 months
  It is for idiopathic membranous nephropathy group. It was calculated according to ckD-EPI 2009 formula

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Xiyuan hospital， China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Fujian Provincial People's Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Henan University of traditional Chinese Medicine, Zhengzhou, Henan
  - Hubei Provincial Hospital of Traditional Chinese Medicine, Wuhan, Hubei
  - Yichang Hospital of Traditional Chinese Medicine, Wuhan, Hubei
  - Affiliated Hospital of Jiangxi University of traditional Chinese Medicine, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No